CLINICAL TRIAL: NCT00484445
Title: Transfer to Another Health Care Facility Following Critical Illness
Status: Completed | Type: Observational
Sponsor: University of Chicago (Other)
Collaborators: The John A. Hartford Foundation (Other); American College of Chest Physicians (Other); Association of Subspecialty Professors (Other)
Responsible Party: Sponsor
Other Study IDs: 12093B
Record Dates: First submitted 2007-06-08; First posted 2007-06-11 (Estimated); Last update posted 2013-09-05 (Estimated); Status verified 2013-09

CONDITIONS: Transfer to a Health Care Facility After Critical Illness
Keywords: Chronic critical illness; Functional status; Outcomes; Post-ICU

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to identify acute and chronic medical conditions that are identifiable early in the course of critical illness that are associated with transfer to another health care facility (versus to home) upon hospital discharge.

DETAILED DESCRIPTION:
Many patients who survive critical illness are unable to return home upon hospital discharge and require prolonged or permanent care in other health care facilities. It would be useful to clinicians, researchers, patients, and patients' families to be able to identify early in the course of critical illness those patients who are at increased risk for this outcome. Currently, few data exist regarding the risk factors for this outcome. This study examines a cohort of survivors of critical illness to identify factors associated with transfer to another health care facility upon hospital discharge.

ELIGIBILITY:
Inclusion Criteria:

* Admission to the University of Chicago Medical Intensive Care Unit during the following periods: July 1997 to February 1998, November/December 2001, and March/April 2002.

Exclusion Criteria:

* Death during the index hospitalization.
* Residence in another health care facility 2 weeks prior to admission.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to an urban medical intensive care unit.
Sampling Method: Probability Sample
Enrollment: 548 (Actual)
Dates: Start 2003-01; Primary Completion 2003-01 (Actual); Study Completion 2003-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian K Gehlbach, MD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago Hospitals, Chicago, Illinois, United States